CLINICAL TRIAL: NCT03930537
Title: DIfference of Femoral Intramedullar Pressure After Implantation of Cemented Versus Non-cemented Femoral Component of Hip Prothesis
Brief Title: Change of Intramedullar Pressure After Implantation of Hip Prothesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Principal Investigator, Skender Ukaj, Specialist of Orthopaedics and Trauma, University Clinical Centre of Kosova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10/2019
Record Dates: First submitted 2019-04-07; First posted 2019-04-29 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Arthroplasty Complications
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip replacement with cemented femoral component (Active Comparator): A special device that measure the pressure will be used to measure the change of pressure before, during and after implantation of cemented femoral component of hip prothesis.
  Interventions: Device: Hip replacement
- Hip replacement with non-cemented femoral component (Active Comparator): A special device that measure the pressure will be used to measure the change of pressure before, during and after implantation of non-cemented femoral component of hip prothesis.
  Interventions: Device: Hip replacement

INTERVENTIONS:
Device: Hip replacement — The hip replacement surgery is when a damaged hip is replaced with artificial one

SUMMARY:
It is well known that the changes in intramedullary canal during orthopedic surgeries can cause variuos complication. The change of femoral intramedullary pressure after implantation of hip replacement and its possible complications are not well studied and the investigators are aiming to give more answer to this issue.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing hip replacement with cemented and non-cemented femoral component

Exclusion Criteria:

* ASA IV
* Patient with periprosthetic fractures
* Patient with hip replacement revision

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-17 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change of pressure in femoral intramedullary canal after implantation of femoral component | The femoral intramedullary pressure will be measured before the cut of femoral neck and continuously during first 10 minutes after the implantation of cemented femoral component
  The pressure in intramedullary canal will be measured with customized device

SECONDARY OUTCOMES:
Difference of arterial pressure after implantation of femoral component | The changes will be measured before implantation and during first 10 minutes after implantation
  The changes will be measured by the device monitor connected to patient
Difference of changes of Leukocyte formula after implantation of femoral component | The blood will be taken from patience 1 hour before and POD1
  The changes will be measured from the blood taken from operated patients
Difference of SpO2 after implantation of femoral component | The changes will be measured before implantation and during first 10 minutes after implantation
  The changes will be measured by the device monitor connected to patient
Difference of SpCO after implantation of femoral component | The changes will be measured before implantation and during first 10 minutes after implantation
  The changes will be measured by the device monitor connected to patient
Difference of changes of CRP after implantation of femoral component | The blood will be taken from patience 1 hour before and POD1
  The changes will be measured from the blood taken from operated patients
Difference of changes of Histamine after implantation of femoral component | The blood will be taken from patience 1 hour before and POD1
  The changes will be measured from the blood taken from operated patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Kosovo, Pristina, Kosovo

REFERENCES:
- [Derived] Ukaj S, Ukaj D, Dervishaj F, Dyla D, Krasniqi E, Elezi G, Obertinca R, Boshnjaku A. Systemic inflammatory response to cemented and uncemented total hip arthroplasty with PMMA bone cement. Sci Rep. 2025 Nov 20;15(1):40957. doi: 10.1038/s41598-025-24695-0. PMID 41266408
- [Derived] Ukaj S, Veslko M, Krasniqi S, Podvorica V, Ukaj F, Ahmeti A, Hernigou P, Cimerman M. Cemented stems in healthy elderly patients result in higher hypoxia despite a paradoxical lower femoral increase of intramedullary pressure. Int Orthop. 2021 Apr;45(4):915-922. doi: 10.1007/s00264-021-04955-0. Epub 2021 Feb 2. PMID 33528632